CLINICAL TRIAL: NCT05050136
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Volixibat in the Treatment of Cholestatic Pruritus in Patients With Primary Biliary Cholangitis
Brief Title: A Study to Evaluate Efficacy and Safety of an Investigational Drug Named Volixibat in Patients With Itching Caused by Primary Biliary Cholangitis
Acronym: VANTAGE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mirum Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VLX-601
Record Dates: First submitted 2021-09-09; First posted 2021-09-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis; PBC
Keywords: Pruritus; PBC; Itching; Cholangitis; Primary Biliary Cholangitis; Hepatobiliary disorders
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Pruritus; Cholangitis; Digestive System Diseases | interventions — volixibat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 Arm 1: Volixibat 20mg (Experimental): Participants randomized to this arm will receive volixibat 20mg twice daily.
  Interventions: Drug: Volixibat
- Part 1 Arm 2: Volixibat 80mg (Experimental): Participants randomized to this arm will receive volixibat 80mg twice daily.
  Interventions: Drug: Volixibat
- Part 1 Arm 3: Placebo (Placebo Comparator): Participants in this arm will receive capsules matched to the study drug minus the active volixibat substance, twice daily.
  Interventions: Drug: Placebo
- Part 2 Arm 1: Volixibat Selected Dose 20mg (Experimental): Participants randomized to this arm will receive volixibat 20mg twice daily.
  Interventions: Drug: Volixibat
- Part 2 Arm 2: Placebo (Placebo Comparator): Participants in this arm will receive capsules matched to the study drug minus the active volixibat substance, twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Volixibat — Oral capsules, administered twice daily. Volixibat is an Ileal Bile Acid Transporter (IBAT) inhibitor.
  Other Names: SHP626
  Arms: Part 1 Arm 1: Volixibat 20mg; Part 1 Arm 2: Volixibat 80mg; Part 2 Arm 1: Volixibat Selected Dose 20mg
Drug: Placebo — Capsules matched to study drug without the active pharmaceutical ingredient
  Arms: Part 1 Arm 3: Placebo; Part 2 Arm 2: Placebo

SUMMARY:
The purpose of this clinical research study is to learn more about the use of the study medicine, volixibat, for the treatment of pruritus (itching) associated with Primary Biliary Cholangitis (PBC), and to assess the possible impact on the disease progression of PBC.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed informed consent at the screening visit as well as comply with all study visits and requirements through the end of the study
* Male or female, age ≥18 years at the screening visit
* Confirmed diagnosis of PBC in line with the AASLD guidelines
* UDCA, anti-pruritic medication and PPAR agonist use will be allowed if meeting additional criteria
* Qualified pruritus associated with PBC as assessed by Adult ItchRO

Exclusion Criteria:

* Pruritus associated with an etiology other than PBC
* Evidence or clinical suspicion of decompensated cirrhosis or a history of decompensation events
* Current symptomatic cholelithiasis or inflammatory gallbladder disease
* History of small bowel surgery/resection impacting the terminal ileum that may disrupt the enterohepatic circulation.
* Evidence, history, or suspicion of other liver diseases; PBC patients with AIH are not excluded
* History of Liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-09-22 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Mean change in the daily itch scores using the Adult Itch Reported Outcome (Adult ItchRO) questionnaire | Baseline to week 28
  The Adult ItchRO is an 11-point NRS measurement of itch severity ranging from 0=no itch to 10=worst possible itch.

SECONDARY OUTCOMES:
Proportion of participants with itch response using the Adult ItchRO | Baseline to week 28
Incidence of adverse events | Baseline to week 28
Changes in alkaline phosphatase | Baseline to week 28
Changes in total bilirubin | Baseline to week 28
Changes in serum bile acid levels | Baseline to week 28
Change in Primary Biliary Cholangitis Quality of Life Measure (PBC-40) | Baseline to week 28
  PBC-40 questionnaire is scored on a scale of 40 to 200, with higher scores indicating poorer quality of life
Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) fatigue questionnaire | Baseline to week 28
  The PROMIS® Fatigue questionnaire is a 5-point response scale. Respondents endorse each item using a 5-point response scale: Never, Rarely, Sometimes, Often, and Always.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS®) sleep disturbance questionnaire | Baseline to week 28
  The PROMIS® Sleep Disturbance in an 8-item measure that assesses quality of sleep, sleep depth, and restoration associated with sleep. It is a 5-point response scale, the specific response options vary by items. The first 4 items use response options that range from Not at all to Very much. The next 3 items use response options that range from Never to Always. The final item assesses sleep quality ranging from Very poor to Very good.

CONTACTS AND LOCATIONS:
Locations (115):
- United States (38):
  - Southern California Research Center, Coronado, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UC Davis, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - Yale University Digestive Diseases, New Haven, Connecticut
  - Covenant Metabolic Specialists, Fort Myers, Florida
  - UF Hepatology Research at CTRB, Gainesville, Florida
  - UF Health Gastroenterology- Emerson, Jacksonville, Florida
  - IHS Health, Kissimmee, Florida
  - Schiff Center for Liver Diseases, Miami, Florida
  - Advanced Research Institute, Inc, New Port Richey, Florida
  - Covenant Research and Clinics, LLC, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Southeast Clinical Research Center, Dalton, Georgia
  - Northwestern University, Chicago, Illinois
  - Loyola University Health System - Loyola Outpatient Center, Maywood, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Ochsner Clinic Foundation-Baton Rouge, Baton Rouge, Louisiana
  - LSU Health Science Center Shreveport, Shreveport, Louisiana
  - Beth Israel Deaconess, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Jackson Liver and GI Specialists, Jackson, Mississippi
  - CHI Health Clinic (Alegent Creighton Clinic)- Gastroenterology-Bergan, Omaha, Nebraska
  - Science 37, Inc (Remote-homebased Telemedicine), Morrisville, North Carolina
  - Cleveland Clinic - Main Campus, Cleveland, Ohio
  - Einstein Healthcare Network - Einstein Medical Center, Philadelphia, Pennsylvania
  - Methodist Le Bonheur Healthcare, Memphis, Tennessee
  - Galen Medical Group, P.C, Tennessee City, Tennessee
  - Amel Med LLC, Austin, Texas
  - Soma Clinical Trials, Denison, Texas
  - Baylor College of Medicine, Houston, Texas
  - Liver Associates of Texas, Houston, Texas
  - Velocity Clinical Research, Waco, Texas
  - University of Utah Health Care, Salt Lake City, Utah
  - MedStar Health Research Institute, Fairfax, Virginia
  - Bon Secours Liver Institute of Hampton Roads Mary Immaculate Hospital, Newport News, Virginia
  - Bon Secours Richmond Community Hospital LLC d/b/a Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Liver Institute Northwest, Seattle, Washington
- Argentina (3):
  - Hospital de Alta Complejidad En Red El Cruce, San Juan Bautista, Buenos Aires
  - Hospital Provincial Del Centenario, Rosario, Santa Fe Province
  - Glenny Corp S.A, CABA
- Belgium (3):
  - Universitair Ziekenhuis Antwerpe UZA, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
- Brazil (5):
  - Centro de Pesquisa Clínica da Bahiana Saúde, Salvador, Estado de Bahia
  - Hospital Das Clínicas Da Ufg, Goiânia, Goiás
  - Centro de Pesquisas Clínicas do HC/UFMG-EBSERH, Belo Horizonte, Minas Gerais
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundação Oswaldo Ramos, São Paulo
- Canada (6):
  - Gordon and Leslie Diamond Health Care Centre, Division of Gastroenterology, Vancouver, British Columbia
  - (G.I.R.I.) GI Research Institute Foundation, Vancouver, British Columbia
  - McMaster University Medical Center, Hamilton, Ontario
  - University Hospital, LHSC, London, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - University of Alberta, Edmonton
- China (7):
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Youan Hospital, Capital Medical University, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Sir Run Run Shaw Hospital -Zhejiang University School of Medicine, Hangzhou
- France (6):
  - CHU Grenoble - Hôpital MICHALLON, Grenoble
  - Hopital Claude Huriez-Digestive system disease clinic, Lille
  - CHU de NICE- Hospital L'Archet 2, Nice
  - Hospital Saint Antoine, Paris
  - Nouvel Hospital Civil, Strasbourg
  - Hospital Paul Brousse- APHP, Villejuif
- Germany (8):
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitätsklinikum Frankfurt am Main, Frankfurt
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Onkologie, Gastroenterologie, Hepatologie und Pneumologie, Leipzig
  - University Hospital Munster, Münster
  - University Hospital Tübingen Medical clinic, Tübingen
  - St. Josefs-Hospital Wiesbaden, Wiesbaden
- Israel (9):
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center - Ein Karem, Liver Institute Kiryat Hadassah POB 12000, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (9):
  - Universita Politecnica delle Marche- Ospedali Riuniti, Ancona
  - ASST Papa Giovanni XXIII, Bergamo
  - Fondazione Ca Granda, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Azienda Ospedale-Università di Padova, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero Universitaria Pisana (AOUP), Pisa
  - Istituto Clinico Humanitas, Rozzano
- Japan (5):
  - National Hospital Organization Nagasaki Medical Center, Ōmura, Nagasaki
  - Ehime University Hospital, Ehime
  - Teine Keijinkai Hospital, Hokkaido
  - Osaka Rosai Hospital, Osaka
  - Toranomon Hospital, Tokyo
- Netherlands (3):
  - Amstedam University Medical Centers, Amsterdam
  - Radboudumc, Nijmegen
  - Erasmus medical center, Rotterdam
- Spain (6):
  - Hospital Universitari Vall d' Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Parc Tauli, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (2):
  - Ente Ospedaliero Cantonale, Lugano
  - University Hospital Zurich(USZ), Zurich
- United Kingdom (5):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Belfast Health & Social Care Trust (BHSCT) Royal Victoria Hospital, Belfast
  - Royal Free Hospital NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - Nottingham University Hospitals NHS Trust, Nottingham

REFERENCES:
- [Derived] Klatzkow H, Bhavsar-Burke I, Pearson M, Wentworth BJ. Primary Biliary Cholangitis in 2025: A New Frontier. Am J Gastroenterol. 2025 Dec 1;120(12):2746-2749. doi: 10.14309/ajg.0000000000003559. Epub 2025 May 29. No abstract available. PMID 40439725